CLINICAL TRIAL: NCT02481635
Title: A Phase I/II Study Evaluating the Feasibility and Safety of Neoadjuvant Gemcitabine/Nab-paclitaxel (GA) and Concurrent Gemcitabine and Radiation Therapy Followed By Pancreatic Resection and Major Arterial Resection for Adenocarcinoma of the Pancreas (ARCAP) in Patients With Advanced Disease
Brief Title: A Study of Gemcitabine/Nab-paclitaxel and Radiation Therapy Followed by Surgery in Patients With Advanced Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARCAP-GA
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer
Keywords: Blood Vessels; Reconstructive Surgery
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine/Nab-paclitaxel, Radiation and Surgery (Experimental): Gemcitabine (neoadjuvant and adjuvant), intravenously, at a dose of 1000 mg/m2 given over 30-40 minutes, on Day 1 of every 28 day cycle for 2 cycles.
  Nab-paclitaxel, intravenously, at a dose of 125 mg/m2 given over 30-40 minutes, on Days 1, 8, and 15 of every 28 day cycle for 2 cycles.
  Radiation Therapy: 50.4 Gy in 28 fractions (1.8 Gy/fraction)
  Surgery: Tumor resection and arterial resection/reconstruction
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Radiation: Radiation Therapy; Procedure: Surgical Resection

INTERVENTIONS:
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Nab-paclitaxel
  Other Names: Abraxane
Radiation: Radiation Therapy
Procedure: Surgical Resection

SUMMARY:
This is a phase 1 (the first phase in testing a new drug, to see how safe a new drug or new indication/population ) and phase 2 (the second phase in testing a new drug or new indication/population to see how effective the drug is) study of neoadjuvant (treatment before the main treatment) with gemcitabine and nab-paclitaxel (abraxane) and gemcitabine and radiation therapy before surgery and then gemcitabine and nab-paclitaxel after surgery in patients with pancreatic cancer that has grown to involve one of the major artery branches.

DETAILED DESCRIPTION:
Gemcitabine and nab-paclitaxel are chemotherapy drugs that are currently approved by Health Canada for use in combination for the treatment of pancreatic cancer. However, the combination of gemcitabine and nab-paclitaxel as a neoadjuvant treatment prior to gemcitabine and radiation is experimental. Surgery to remove or reconstruct the major artery is also experimental.

ELIGIBILITY:
Inclusion Criteria:

Surgical:

* Medically fit for major pancreatic surgery
* No evidence of metastases
* No prior resection
* Arterial involvement limited to a single major vessel and is resectable
* Tumour-free margins could be achieved
* Acceptable length of vessel
* Mass considered otherwise resectable by current standards

General:

* Less than 70 years old
* Performance status <=2
* Has pancreatic adenocarcinoma
* Adequate bone marrow and organ function
* Therapeutic heparin is allowed
* Taking chronic erythropoietin are permitted
* Not pregnant
* Agree to use contraception
* Able to provide written consent

Exclusion Criteria:

Surgical:

* Aortic involvement
* Involvement of 2 major arterial trunks
* SMV/portal venous occlusion, cannot be reconstructed
* Extensive venous involvement, no arterial involvement
* Disease progression on neo-adjuvant treatme

General:

* Concurrent cancer diagnosis
* Other malignancies unless all therapy completed, no disease for >=3 years
* Prior radiotherapy or chemo within 1 year, to pancreas
* Bone marrow transplant/stem cell rescue
* Major surgery <4 wks prior
* Distant metastases
* Renal dysfunction
* Pulmonary insufficiency
* History of cardiac disease
* Active systemic infection(s) or any other related illnesses
* Known HIV, HBV, HCV
* History of solid organ transplant, cardiovascular disease, inflammatory bowel disease, or underlying neuropathy
* Conditions interfering with patient participation
* Known or suspected allergy to study drugs
* Pregnant or breast-feeding
* Therapeutic coumadin
* More than or equal to Grade 2 pre-exiting peripheral neuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2024-12-10 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Type and the severity of side effects | 5 years

SECONDARY OUTCOMES:
Number of surviving patients at 1 year after treatment | 1 year
Number of patients who disease has not progressed | 2 years
Number of patients that are able to receive surgery after chemoradiation | 5 years
Average length of hospital stay per patient | 5 years
Number of surviving patients at 30-days after surgery | 30 days after surgery
Number of surviving patients at 90-days after surgery | 90 days after surgery
Number of patients who need to be re-admitted to the hospital at 90-days after surgery | 90 days after surgery
Time to Progression | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Neesha Dhani, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada